CLINICAL TRIAL: NCT05051436
Title: The Effects of Mirabegron and Tadalafil on Glucose Tolerance in Prediabetics
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Philip Kern (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Philip Kern, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 55665; R01DK128033 (NIH)
Record Dates: First submitted 2021-09-10; First posted 2021-09-21 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Pre-diabetes; Obesity
Keywords: Tadalafil; Mirabegron
MeSH Terms: conditions — Glucose Intolerance; Obesity | interventions — mirabegron; Tadalafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Mirabegron (M) (Experimental): Drug will be administered for 12 weeks after baseline procedures.
  Interventions: Drug: Mirabegron 50 MG
- Tadalafil (T) (Experimental): Drug will be administered for 12 weeks after baseline procedures.
  Interventions: Drug: Tadalafil 10 MG
- Mirabegron and Tadalafil (MT) (Experimental): Both drugs will be administered for 12 weeks after baseline procedures.
  Interventions: Drug: Mirabegron 50 MG; Drug: Tadalafil 10 MG
- Placebo (P) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mirabegron 50 MG — Mirabegron 50 mg/day will be administered for 14 weeks.
  Arms: Mirabegron (M); Mirabegron and Tadalafil (MT)
Drug: Tadalafil 10 MG — Tadalafil 10 mg/day will be administered for 14 weeks after baseline procedures.
  Arms: Mirabegron and Tadalafil (MT); Tadalafil (T)
Drug: Placebo — Placebo will be administered for 14 weeks after baseline procedures.
  Arms: Placebo (P)

SUMMARY:
The investigator hypothesizes that treatment with the ß3 agonist mirabegron results in improved glucose metabolism, including a reversal of prediabetes in obese, insulin-resistant human research participants, and this is further improved by combination therapy with tadalafil. The investigator will comprehensively analyze glucose homeostasis in prediabetic patients treated for 14 weeks with mirabegron, tadalafil or both drugs as compared to a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Hemoglobin A1C between 5.7 and 6.4
* Body mass index between 27 and 45

Exclusion Criteria:

* Diabetes
* Chronic use of any antidiabetic medications
* Any unstable medical condition
* Use of steroids or daily use of NSAIDS
* History of chronic inflammatory conditions
* Use of anticoagulants
* Contraindications to the use of mirabegron or tadalafil
* Any condition deemed risky by the study physician

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2021-12-13 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Oral glucose tolerance test | Baseline
  Participants will complete a standard oral glucose tolerance test using 75 g of glucose at baseline and blood glucose will be measured.
Oral glucose tolerance test | 14 weeks
  Participants will complete a standard oral glucose tolerance test using 75 g of glucose at 14 weeks and blood glucose will be measured.

SECONDARY OUTCOMES:
Hemoglobin A1C | Baseline
  Participant hemoglobin A1C will be evaluated at baseline.
Hemoglobin A1C | 14 weeks
  Participant hemoglobin A1C will be evaluated at 14 weeks.

OTHER OUTCOMES:
Fat biopsy | Baseline
  Beiging of fat as measured in the lab by histochemistry.
Fat biopsy | 14 weeks
  Beiging of fat as measured in the lab by histochemistry.
Muscle biopsy | Baseline
  Fiber type, as measured in the lab by histochemistry.
Muscle biopsy | 14 weeks
  Fiber type, as measured in the lab by histochemistry.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Kern, M.D., Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No